CLINICAL TRIAL: NCT01638325
Title: A Study to Assess the Pharmacokinetics, Glucodynamics, Safety, and Tolerability of Single Subcutaneous Injections of Insulin Lispro With BioChaperone Excipient in Healthy Volunteers
Brief Title: A Study of Insulin Lispro With BioChaperone Excipient in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14771; H9D-MC-ITAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro (Active Comparator): 15 international units (IU) insulin lispro administered once subcutaneously (SC) during 1 of 3 dosing periods. There is a minimum 7 day washout between dosing periods.
  Interventions: Drug: Insulin Lispro
- BC106 Insulin Lispro (Experimental): 15 up to 30 IU BC106 insulin lispro administered once SC during 2 of 3 dosing periods. There is a minimum 7 day washout between dosing periods.
  Interventions: Drug: BC106 insulin lispro

INTERVENTIONS:
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro
Drug: BC106 insulin lispro — Administered SC
  Other Names: BioChaperone insulin lispro
  Arms: BC106 Insulin Lispro

SUMMARY:
BC106 is a molecule that when injected with insulin lispro may change the speed of absorption of insulin lispro. The purpose of this study will be to evaluate the safety of BC106 insulin lispro and any side effects that might be associated with it, blood levels of insulin lispro after injection under the skin and how BC106 insulin lispro affects blood sugar after injection under the skin. There is a minimum 7 day washout between single doses.

ELIGIBILITY:
Inclusion Criteria:

* Are not of child-bearing potential
* Have a body mass index (BMI) between 18 and 29.9 kilograms per square meter (kg/m^2), inclusive
* Are nonsmokers or have not smoked for at least 6 months prior to entering the study
* Have a fasting plasma glucose less than 6.0 millimoles per liter (mmol/L) at screening

Exclusion Criteria:

* Have known allergies to insulin or its excipients, or related drugs, or history of relevant allergic reactions of any origin including allergies to dextrans
* Have a history of first-degree relatives known to have diabetes mellitus
* Have used systemic glucocorticoids within 3 months prior to entry into the study
* Have donated or had a blood loss of 450 milliliters (mL) 3 months prior to study enrollment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration curve (AUC) | Baseline up to 8 hours post administration of study drug
Pharmacokinetics: Maximum concentration (Cmax) | Baseline up to 8 hours post administration of study drug
Pharmacokinetics: Time of maximum concentration (Tmax) | Baseline up to 8 hours post administration of study drug

SECONDARY OUTCOMES:
Glucodynamic response: Time to maximum infusion rate (tRmax) during euglycemic clamps of BC106 insulin lispro | Baseline up to 30 days
Pharmacokinetics: Within-participant variability of time to maximum drug concentration (tmax) of BC106 insulin lispro | Baseline up to 30 days
Glucodynamic within-participant variability of time to maximum glucose infusion rate (tRmax) for BC106 insulin lispro | Baseline up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore